CLINICAL TRIAL: NCT00447018
Title: Equimolar Doses of Mannitol and Hypertonic Saline in the Treatment of Elevated Intracranial Pressure
Brief Title: Mannitol Versus Hypertonic Saline Solution in the Treatment of Elevated Intracranial Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0224
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Intracranial Hypertension
Keywords: intracranial pressure; mannitol; hypertonic saline solution; brain injury; traumatic brain injury; Adult patients; With elevation of intracranial pressure (ICP > 20 mmHg)
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries; Brain Injuries, Traumatic | interventions — Mannitol; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 20% mannitol
Drug: 7.45% hypertonic saline solution

SUMMARY:
The purpose of this study is to determine whether mannitol is as effective as hypertonic saline solution in the treatment of elevated intracranial pressure in patients with brain injury.

DETAILED DESCRIPTION:
Elevation of intracranial pressure (ICP) to more than 20 mmHg plays a major role in the worsening of the neurological status through the impairment of brain perfusion. In an effort to reduce the intensity and the time spent with increased ICP, infusion of mannitol has been the recommended first-line agent for years. The growing interest in the use of hypertonic saline solutions (HSS) in this clinical setting has, however, challenged the use of mannitol. Because mannitol and HSS may differ regarding their clinically relevant mechanisms of action, there is a need to determine which osmotic compound could be the most appropriate in patients with elevated ICP. We conduct thus a parallel, randomized controlled trial comparing the effects of an equimolar infusion of 20% mannitol or 7.45% HSS without colloid in patients with elevated ICP. The primary end point of this trial is the magnitude of ICP and of cerebral perfusion pressure (CPP) changes following treatment during a study period of 120 min.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* sustained elevated intracranial pressure to more than 20 mmHg for more than 10 min
* mechanically ventilated in stable conditions for more than 2 hours prior to the study
* serum osmolality ranged between 280 and 320 mOsm/kg

Exclusion Criteria:

* imminent cranial or extracranial surgery
* leakage or drainage of cerebral spinal fluid
* unstable respiratory and hemodynamic conditions
* oliguric renal failure
* anemia
* use of mannitol or HSS in the previous 6 hours
* concomitant use of thiopentone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-10; Study Completion 2005-06

PRIMARY OUTCOMES:
Magnitude of ICP and of cerebral perfusion pressure (CPP) changes following osmotherapy during a study period of 120 min.

SECONDARY OUTCOMES:
Effects of treatment on blood flow velocities (FV) of middle cerebral artery using continuous transcranial doppler.
Effects of treatment on brain oxygenation using brain tissue oxygen tension (PbrO2) probe.
Effects of treatment on biochemical data (serum sodium and osmolality, urine output).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Payen, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Hopital Michallon, Grenoble, France

REFERENCES:
- [Result] Battison C, Andrews PJ, Graham C, Petty T. Randomized, controlled trial on the effect of a 20% mannitol solution and a 7.5% saline/6% dextran solution on increased intracranial pressure after brain injury. Crit Care Med. 2005 Jan;33(1):196-202; discussion 257-8. doi: 10.1097/01.ccm.0000150269.65485.a6. PMID 15644669
- [Result] Vialet R, Albanese J, Thomachot L, Antonini F, Bourgouin A, Alliez B, Martin C. Isovolume hypertonic solutes (sodium chloride or mannitol) in the treatment of refractory posttraumatic intracranial hypertension: 2 mL/kg 7.5% saline is more effective than 2 mL/kg 20% mannitol. Crit Care Med. 2003 Jun;31(6):1683-7. doi: 10.1097/01.CCM.0000063268.91710.DF. PMID 12794404